CLINICAL TRIAL: NCT05982197
Title: The Effect of Curcuma Long Oral Gel in Relation to Salivary Epidermal Growth Factor & Interleukin-8 on Radiation Induced Oral Mucositis in Iraqi Cancer Patients
Brief Title: Curcumin Gel On Radiation Induced Oral Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, sarah adnan abdul-jabbar, principal investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 705722
Record Dates: First submitted 2023-06-22; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Radiation-Induced Mucositis; Head and Neck Cancer
Keywords: Radiation induced oral mucositis; Head and neck cancer; Curcuma longa; EGF; IL8
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Reference Standards

STUDY DESIGN:
Intervention Model Description: Two groups A) curcuma longa oral gel group B) standard treatment group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Curcuma longa oral gel group (Active Comparator)
  Interventions: Drug: Curcumin Gel
- Standard treatment group (Active Comparator)
  Interventions: Drug: Standard Preparation

INTERVENTIONS:
Drug: Curcumin Gel — Curcuma longa oral gel for prevention radiation induced oral mucositis
  Arms: Curcuma longa oral gel group
Drug: Standard Preparation — Standard preparation for prevention radiation induced oral mucositis
  Arms: Standard treatment group

SUMMARY:
The goal of this clinical study is to investigate the effect of a curcuma longa oral gel (curenext) on reducing radiation-induced oral mucositis severity in cancer patients and provide a context for understanding if there is a relationship between the curcumin clinical effect and production of EGFs and IL8.

Researchers will compare between curcumin group and standard treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 16 years having histopathologically confirmed cancer in head and neck region who planned to have radiation with head and neck mask.
* Scheduled for 6-8 weeks of radiotherapy with 60-70Gy radiation (200cgy/fraction for 5 days/week).

Exclusion Criteria:

* patient with hodgkin lymphoma.
* Any allergy to curcumin or other condiments.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-07-02 (Actual)

PRIMARY OUTCOMES:
Onset of radiation induced mucositis | Assessment every week starting from first visit until the onset of mucositis (up to 2 months)
  Onset (at which week) of radiation induced mucositis in relation to EGF and IL8
Change in severity of radiation induced mucositis | Assessment every week starting from first visit of radiation unit it completion (average of 2 months)
  Change in severity (degree of illness) of radiation induced mucositis in relation to EGF & IL-8 by World Health Organization (WHO) mucositis scale {0: no. 1: mild. 2 and 3 : moderate. 4: severe}

CONTACTS AND LOCATIONS:
Locations (1):
- Nuclear medicine and radiation therapy hospital, Baghdad, Iraq